CLINICAL TRIAL: NCT00310778
Title: Effects of Sodium Intake on Pharmacokinetic/Pharmacodynamic Relationship of a Single Dose of a Renin Angiotensin System-Blocker, or a Beta-Blocker in Normotensive Sodium-Depleted or Replated Volunteers in a Cross-Over Study
Brief Title: Effects of Sodium Intake on (PK/PD) Relationship of a Single Dose of a Renin Angiotensin System-Blocker
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle Brindel, Department Clinical Research of Developpement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P051201
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Healthy
Keywords: High sodium diet; Low sodium diet; Renin-angiotensin system blockers; AT1 receptor (AT1R) antagonist; ACE inhibition
MeSH Terms: interventions — Diet, Sodium-Restricted; Ramipril; Valsartan; candesartan; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): treatment
  Interventions: Drug: high sodium diet; Drug: low sodium diet; Drug: ramipril 10 mg; Drug: valsartan 160 mg; Drug: candesartan 8 mg; Drug: atenolol 50 mg

INTERVENTIONS:
Drug: high sodium diet — high sodium diet
Drug: low sodium diet — low sodium diet
Drug: ramipril 10 mg — ramipril 10 mg
Drug: valsartan 160 mg — valsartan 160 mg
Drug: candesartan 8 mg — candesartan 8 mg
Drug: atenolol 50 mg — atenolol 50 mg

SUMMARY:
The impact of sodium intake on plasma drug concentrations has previously been reported in the literature for verapamil and quinidine but, to the investigators' knowledge, never with renin-angiotensin system blockers such as AT1R antagonists and angiotensin converting enzyme inhibitors.

DETAILED DESCRIPTION:
The impact of sodium intake on plasma drug concentrations concentrations obtained after a single oral dose of RAS blocking drugs (ramipril 10 mg, valsartan 160 mg, candesartan 8 mg) or a blocker as control (ATENOLOL 50 mg) will be compared in healthy normotensive men randomly assigned to a 6-day replated-sodium diet or a sodium depletion.

ELIGIBILITY:
Inclusion Criteria:

* 64 (16 per treatment goup) non-smoking healthy male volunteers
* Aged between 18 and 35 years after a complete clinical examination
* Safety laboratory measurements
* Having given written informed consent.

Exclusion Criteria:

* hypertension
* known disease
* diabetes mellitus
* known hypersensitivity
* contraindication to ACE inhibitors
* history of cardiac or pulmonary disease or asthma conditions which do not permit medical follow-up and compliance with the study protocol.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) up to the 48 hour time point of plasma drug concentrations between a replated-sodium diet and sodium depletion | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michel Azizi, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre d'Investigation Clinique 9201 Hôpital Européen Georges Pompidou, Paris, France

REFERENCES:
- [Background] Azizi M, Menard J, Bissery A, Guyenne TT, Bura-Riviere A, Vaidyanathan S, Camisasca RP. Pharmacologic demonstration of the synergistic effects of a combination of the renin inhibitor aliskiren and the AT1 receptor antagonist valsartan on the angiotensin II-renin feedback interruption. J Am Soc Nephrol. 2004 Dec;15(12):3126-33. doi: 10.1097/01.ASN.0000146686.35541.29. PMID 15579516